CLINICAL TRIAL: NCT07404696
Title: Early Interceptive (Headgear-Activator, Twin Block, Invisalign MA) Versus Later Fixed Appliance Treatment in Class II Malocclusion: A Randomized Clinical Trial
Brief Title: Comparison of Early Interceptive Orthodontic Appliances (Traditional and Novel) and Later Fixed Appliance Treatment in Class II Malocclusion.
Acronym: MACTWin
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Västra Götalandsregionen (Other); Region Halland (Other); Göteborg University (Other)
Responsible Party: Principal Investigator, Anna Westerlund, Professor, Göteborg University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCT: Comparing Class II TX
Record Dates: First submitted 2025-12-17; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Class II Malocclusion; Class II Malocclusion, Division 1; Overjet
MeSH Terms: conditions — Overbite; Malocclusion, Angle Class II | interventions — Orthodontic Appliances, Fixed

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled, investigator-blinded, multicentre clinical trial.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Head gear activator (Experimental): Treatment with head gear activator orthodontic appliance.
  Interventions: Device: Head gear activator
- Twin Block (Experimental): Treatment with Twin Block appliance
  Interventions: Device: Twin Block
- Invisalign Mandibular Advancement (Experimental): Treatment with Invisalign mandibular advancement featuring occlusal blocks.
  Interventions: Device: Invisalign mandibular advancement
- Fixed appliance (Experimental): Participants will serve as an observation (no treatment) control group during the trial period for 18 months. After completion of the observation phase, they will receive orthodontic treatment with fixed appliances. Outcomes from this delayed intervention will be compared with the three early intervention groups.
  Interventions: Device: Fixed appliance

INTERVENTIONS:
Device: Head gear activator — Activator with extra orala head gear traction
  Arms: Head gear activator
Device: Twin Block — Twin Block orthodontic appliance
  Arms: Twin Block
Device: Invisalign mandibular advancement — Invisalign mandibular advancement featuring occlusal blocks
  Arms: Invisalign Mandibular Advancement
Device: Fixed appliance — Fixed appliance in upper and lower jaw
  Arms: Fixed appliance

SUMMARY:
Background Approximately 15% of children have a Class II malocclusion, where the maxilla is positioned anterior to the mandible, and around 90% of these children also present with an increased overjet. Increased overjet is associated with a higher risk of dental trauma and psychosocial consequences such as bullying and reduced oral health-related quality of life (OHRQoL).

Functional orthodontic appliances (e.g., headgear-activator and Twin-block) have long been used to reduce overjet through dentoalveolar effects and by influencing mandibular position and growth. More recently, digital solutions such as Invisalign's mandibular advancement appliance have been introduced, with potential advantages including improved wear time and simultaneous tooth alignment. However, there is currently limited evidence regarding treatment outcomes, patient experience, and cost-effectiveness of these newer appliances compared with established functional appliances.

Aim The primary aim is to compare treatment outcomes, patient experience, and cost-effectiveness of interceptive orthodontic treatment using three different appliances. The overall aim is to determine whether interceptive treatment of Class II malocclusion with large overjet is effective, and if so, which interceptive modality should be preferred.

Study design and setting

A total of 144 patients aged 9-13 years with Class II malocclusion and large overjet will be randomized into four groups:

* Headgear-activator
* Twin-block
* Aligner Mandibular advancement
* Control

Participants will be treated at four Orthodontic Specialist Clinics within the National Health Service in Region Halland and Västra Götaland, Sweden. Treatments will be provided by two experienced orthodontic specialists.

Follow-up and data collection

Clinical examinations will be performed at:

* Baseline (T0)
* 9 months into treatment (T1)
* End of treatment (T2) Appliance checks will occur every 8 weeks. Digital scans of the occlusion will be collected at T0, T1, and T2. Lateral cephalometric radiographs will be taken at T0 and T2.

Outcomes and planned analyses

The trial will generate three studies with distinct outcomes:

1. Treatment outcomes Primary outcome: dental treatment effectiveness measured as overjet reduction. Secondary outcomes: other dental variables, skeletal outcomes, and extraoral outcomes.
2. Patient-reported outcomes

   All treated patients will complete two digital questionnaires:
   * Child Perception Questionnaire (CPQ): assesses the child's perception of their teeth before and after treatment.
   * Orthodontic Treatment Impact Questionnaire (OTIQ): assesses the child's experience of orthodontic treatment and the appliance.

   These outcomes will be used to evaluate changes in OHRQoL from pre- to post-treatment and to compare experiences across treatment modalities.
3. Cost-effectiveness analysis The economic evaluation will include direct, indirect, and societal costs. Treatment duration, number and length of appointments, and cancellations/no-shows will be recorded.

   * Direct costs: premises, staff salaries, materials, and laboratory costs.
   * Indirect costs: parental loss of income due to absence from work.
   * Societal costs: direct + indirect costs. Costs will be related to treatment outcomes to estimate cost-effectiveness across the treatment arms.

Additional comparison: early vs late treatment Furthermore, after completing 18 months the control group, and half of the functional appliance patients will receive treatment with fixed appliances. This enables an additional comparison of early interceptive treatment versus later treatment using the same outcomes: treatment effectiveness, patient-reported outcomes, and cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Children age 9-13 years at the start of the trial
* Mixed dentition, DS3M1
* Excessive overjet ≥6 mm
* First permanent molars in at least half cusp Cl II relation bilaterally
* Incomplete lip closure

Exclusion Criteria:

* Treatment needing extractions due to severe crowding
* Earlier orthodontic treatment
* Mouth breathing
* Ongoing sucking habits
* Syndromic patients

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 144 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2031-03-01 (Estimated); Study Completion 2031-03-01 (Estimated)

PRIMARY OUTCOMES:
Part I: Dental treatment result: Overjet reduction | 18 months
  Change in dental overjet compared to baseline. Unit: millimetres (mm). Direction of effect: Lower post-treatment overjet (i.e. greater reduction from baseline) indicates a better outcome; higher overjet values indicate a worse outcome.

SECONDARY OUTCOMES:
Part I: Dental treatment result: Sagittal relation, overbite | 18 months
  Sagittal relationship at the end of treatment, evaluated by both molar and canine relationships. Unit: millimetres (mm).
  Direction of effect:
  Change towards Class I in molar and canine relation compared with baseline is favorable.

OTHER OUTCOMES:
Part I: Basal treatment result | 18 months
  Skeletal treatment outcomes will be evaluated as changes in SNA, SNB, ANB, NL/ML, Wits, Ils/NL, Ili/ML, Ils/NA, and Ili/NB between baseline and the end of treatment. The measurements will be obtained from lateral cephalometric radiographs. Unit: degrees (°). Direction of effect: Non-linear; mid-range values are favourable, whereas both low and high values are clinically unfavourable.
Part I: Extra oral treatment result | 18 months
  Changes in profile angle and lip closure from before start of the treatment and end of the treatment. The mesurements will be done on standardized photographs. Unit: degrees (°). Direction of effect: Non-linear; mid-range values are favourable, whereas both low and high values are clinically unfavourable.
Part II: Oral Health Related Quality of life (ORHQoL) | 18 months
  Changes in OHRQoL from baseline compared to end of the treatment. Unit: OHRQoL score (higher = worse)
Part II: Patient experience of the orthodontic treatment | 18 months
  The results of the Orthodontic Treatment Impact Questionnaire (OTIQ) will be compared across all groups to evaluate patient experience with the different orthodontic appliances. Score- higher scores reflect more negative impact of treatment
Part III: Direct costs | 18 months
  The difference in direct costs between the different treatment alternatives. Unit: currency units per patient (e.g. EUR per completed treatment) Direction of effect: Lower values indicate lower direct costs (favourable).
Part III: Indirect costs | 18 months
  The difference in indirect costs between the different treatment alternatives. Unit: currency units per patient (e.g. EUR per completed treatment) Direction of effect: Lower values indicate lower direct costs (favourable).
Part I: Societal costs | 18 months
  The difference in societal costs between the treatment alternatives. Societal costs are defined as the sum of direct and indirect costs. Unit: currency units per patient (e.g. EUR per completed treatment) Direction of effect: Lower values indicate lower direct costs (favourable).

CONTACTS AND LOCATIONS:
Overall Officials: Anna Westerlund, Professor, Principal Investigator — Department of Orthodontics, Institution of Odontology, Sahlgrenska Academy, University of Gothenburg
Locations (3):
- Sweden (3):
  - Sahlgrenska Academy, Gothenburg
  - Orthodontic Specialist Clinic, Halmstad
  - Orthodontic Specialist Clinic, Kungsbacka

IPD SHARING:
Plan to Share IPD: Undecided
Charing individual patient data is not approved in the ethical approval.